CLINICAL TRIAL: NCT05926960
Title: A PHASE 2, RANDOMIZED, OPEN-LABEL STUDY OF ENCORAFENIB AND BINIMETINIB PLUS PEMBROLIZUMAB VERSUS NIVOLUMAB AND IPILIMUMAB IN PARTICIPANTS WITH BRAF V600E/K MUTATION-POSITIVE MELANOMA WHO PROGRESSED DURING OR AFTER PRIOR TREATMENT WITH ANTI-PD-1 THERAPY
Brief Title: A Study Comparing 3 Study Medicines (Encorafenib, Binimetinib, Pembrolizumab) to 2 Study Medicines (Ipilimumab and Nivolumab) in Patients With Advanced Melanoma
Acronym: PORTSIDE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4221023; KEYNOTE-C92 (Other: Alias Study Number); 2023-509471-17-00 (Registry Identifier: CTIS (EU)); MK-3475-C92 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-04-03; First posted 2023-07-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: BRAF; BRAF V600E/K melanoma; metastatic melanoma; advanced melanoma; skin cancer; portside
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — encorafenib; binimetinib; pembrolizumab; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Triplet (Experimental): encorafenib and binimetinib in combination with pembrolizumab
  Interventions: Drug: encorafenib; Drug: binimetinib; Drug: pembrolizumab
- Doublet (Active Comparator): ipilimumab and nivolumab
  Interventions: Drug: ipilimumab; Drug: nivolumab

INTERVENTIONS:
Drug: encorafenib — encorafenib
  Other Names: BRAFTOVI
  Arms: Triplet
Drug: binimetinib — binimetinib
  Other Names: MEKTOVI
  Arms: Triplet
Drug: pembrolizumab — pembrolizumab
  Other Names: KEYTRUDA®
  Arms: Triplet
Drug: ipilimumab — ipilimumab
  Other Names: YERVOY
  Arms: Doublet
Drug: nivolumab — nivolumab
  Other Names: OPDIVO
  Arms: Doublet

SUMMARY:
The purpose of this study is to learn about the effects of 3 study medicines (encorafenib, binimetinib, pembrolizumab) compared to 2 study medicines (ipilimumab and nivolumab) given for the treatment of melanoma.

Melanoma is a type of cancer that starts in the cells that give color to your skin.

The study is seeking participants who:

* have advanced or metastatic melanoma (has spread to other parts of the body);
* have a certain abnormal gene called "BRAF".
* have taken nivolumab or pembrolizumab treatment before this study.

Participants will either receive:

* pembrolizumab given by intravenous infusion (directly into a vein) every 3 weeks at the study clinic. Participants will also receive encorafenib and binimetinib by mouth every day at home,
* or will receive ipilimumab and nivolumab given by intravenous infusion (directly into a vein) every 3 weeks at the study clinic 4 times. This will be followed by nivolumab given by intravenous infusion every 4 weeks at the study clinic.

Both pembrolizumab and nivolumab will be given for a maximum of around 2 years. However, there is no time limit for encorafenib and binimetinib treatment.

The study team will see how each participant is doing after receiving the study treatments during regular visits to the study clinic.

DETAILED DESCRIPTION:
The purpose of the study is to compare the efficacy of a triplet therapy (encorafenib, binimetinib, pembrolizumab) versus a doublet/control therapy (nivolumab and ipilimumab). Participants will have metastatic or unresectable locally advanced BRAF V600E/K-mutant melanoma, which progressed during or after prior treatment in the adjuvant or first-line metastatic setting, with an approved anti-PD-1 monotherapy (pembrolizumab or nivolumab),

Approximately 150 participants will be randomized in a 1:1 ratio to the triplet or the doublet/control therapy (75 participants in each arm). Randomization will be stratified by baseline serum LDH level, and by type of PD-1 resistance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 years of age at the time of informed consent.
* Histologically confirmed unresectable (Stage IIIB, IIIC, or IIID) or metastatic (Stage IV) cutaneous melanoma, according to the AJCC 8th edition.
* Documented evidence of a BRAF V600E or V600K mutation.
* Availability of adequate tumor tissue (archival or newly obtained; block or slides) to submit to the sponsor central laboratory(ies) during the screening period for central biomarker analyses .
* Must have received only 1 prior line of systemic therapy for melanoma (either adjuvant therapy or first-line anti-PD-1 monotherapy (ie, nivolumab or pembrolizumab)
* Must have anti-PD-1 resistant disease (primary or secondary) with confirmed disease progression per RECIST v1.1 either during or after receipt of an approved anti-PD-1 monotherapy (ie, nivolumab or pembrolizumab) for melanoma, defined according to the SITC Immunotherapy Resistance Taskforce (Kluger et al, 2020).
* Have at least one measurable lesion per RECIST v1.1.
* ECOG PS of 0-1, and adequate organ and cardiac function, including LVEF ≥50% by cardiac imaging.

Exclusion Criteria:

* Mucosal or ocular melanoma.
* Diagnosis of immunodeficiency or an active autoimmune disease that required systemic treatment with chronic systemic steroid therapy or any other form of immunosuppressive therapy within the past 2 years.
* Clinically significant cardiovascular diseases.
* History of thromboembolic or cerebrovascular events ≤12 weeks prior to randomization.
* History or current evidence of RVO or current risk factors for RVO.
* Concurrent neuromuscular disorder that is associated with the potential of elevated CK.
* Active bacterial, fungal, or viral infection requiring systemic therapeutic treatment within 2 weeks prior to randomization.
* Current non-infectious pneumonitis/interstitial lung disease or history of noninfectious pneumonitis/interstitial lung disease requiring steroids.
* Prior or current symptomatic brain metastasis, leptomeningeal disease or other active CNS metastases.
* Participants who permanently discontinued prior anti-PD-1 therapy due to toxicity or will be unable to tolerate combination therapy based on investigator judgement are excluded.
* Prior treatment with ipilimumab; prior combined immunotherapy blockade with anti-PD-1/L-1; prior treatment with a BRAFi and/or MEKi; or previous administration of an investigational anti-cancer agent for the adjuvant or first-line treatment of melanoma prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) is defined as the proportion of participants in each treatment arm with a confirmed best overall response of either Complete Response (CR) or Partial Response (PR), as determined by investigator assessment per RECIST v1.1 | Time from the date of randomization to the earliest date disease progression, or start of subsequent anticancer therapy, or death due to any cause (assessed up to approximately 48 months).

SECONDARY OUTCOMES:
Progression Free Survival in each treatment arm | Time from the date of randomization to the earliest date of disease progression, as determined by investigator assessment per RECIST v1.1, or death due to any cause, whichever occurs first (assessed up to approximately 48 months)
Overall Survival in each treatment arm | Time from date of randomization to the date of death due to any cause or the last known alive date (assessed up to approximately 48 months)
Duration of Response (CR or PR) in each treatment arm | Time from the date of the first documented response (CR or PR) to the earliest date of disease progression, as determined by investigator assessment per RECIST v1.1, or death due to any cause (assessed up to approximately 48 months)
Disease Control Rate (proportion of participants with a confirmed best overall response of CR, PR or SD) in each treatment arm | Time from the date of randomization to the earliest date of disease progression, or start of subsequent anticancer therapy (assessed up to approximately 48 months)
Time to Response (CR or PR) | Time from the date of randomization to the date of first documented response (CR or PR), as determined by investigator assessment per RECIST v1.1 (assessed up to approximately 48 months)
Progression Free Survival 2 in each treatment arm | Time from date of randomization to date of discontinuation of next-line treatment after 1st disease progression, 2nd disease progression after initiation of next line treatment, or death due to any cause (assessed up to approximately 48 months)
Incidence and severity of Adverse Events (AEs) and changes in clinical laboratory parameters, vital signs, and cardiac assessments. | Time from first dose of study intervention through 28 days after the last dose of study intervention
  Number of participants with treatment emergent Adverse Events as as assessed per National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 4.03).
Patient Reported Outcomes using EORTC QLQ-C30 questionnaires in each treatment arm | Change from Baseline until Progressive Disease, death, withdrawal of consent, lost to follow-up, or end of study, whichever occurs first (assessed up to approximately 48 months)
  EORTC (European Organization for Research and Treatment of Cancer) QLQ-30 includes 5 functional scales (physical, role, emotional, cognitive and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/Quality of Life scale
Patient Reported Outcomes using EuroQOL EQ-5D-5L questionnaires in each treatment arm | Change from Baseline until Progressive Disease, death, withdrawal of consent, lost to follow-up, or end of study, whichever occurs first (assessed up to approximately 48 months)
  The EQ-5D-5L is a standardized measure of health utility that provides a single index value of health status and contains 1 item for each of 5 dimensions of HRQoL (ie, mobility, self-care, usual activities, pain or discomfort, and anxiety or depression).
BRAF V600E/K Variant Allele Frequency and/or overall mean Variant Allele Frequency from circulating tumour DNA analysis in each treatment arm | Change from baseline, Day 1 of Cycle 2 (after 3 weeks), and End of Treatment (assessed up to approximately 48 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- Germany (6):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Fachklinik Hornheide, Münster, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
- Italy (8):
  - Istituto Nazionale Tumori Regina Elena, Rome, ROMA
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Azienda Ospedaliero Universitaria Senese, Siena, Tuscany
  - AO Santa Maria della Misericordia, Perugia, Umbria
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
- Pratia MCM Krakow, Krakow, Poland
- Slovakia (2):
  - Narodny onkologicky ustav, Bratislava
  - Neovizia, s.r.o., Bratislava
- Spain (7):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Catalunya [cataluña]
  - Hospital General Universitario de Valencia, Valencia, Valenciana, Comunitat
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4221023